CLINICAL TRIAL: NCT02631044
Title: A Phase 1, Multicenter, Open-Label Study of JCAR017, CD19-targeted Chimeric Antigen Receptor (CAR) T Cells, for Relapsed and Refractory (R/R) B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Study Evaluating the Safety and Pharmacokinetics of JCAR017 in B-cell Non-Hodgkin Lymphoma (TRANSCEND-NHL-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017001
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Non-Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle-cell Lymphoma; Primary Mediastinal B-cell Lymphoma
Keywords: JCAR017; chimeric antigen receptor; non-Hodgkin lymphoma; CAR; CAR T cells; autologous T cell therapy; cell therapy; NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JCAR017 1-dose schedule (Experimental): Each cycle of JCAR017 (lisocabtagene maraleucel) will be administered as 1 intravenous (IV) injection
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel) single-dose schedule
- JCAR017 2-dose schedule (no longer accruing) (Experimental): Each cycle of JCAR017 (lisocabtagene maraleucel) will be administered as 2 intravenous (IV) injections
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel) 2-dose schedule

INTERVENTIONS:
Biological: JCAR017 (lisocabtagene maraleucel) single-dose schedule — Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JCAR017. During JCAR017 production, participants may receive low-dose chemotherapy for disease control. Upon successful generation of JCAR017 product, participants will receive treatment with JCAR017 therapy. Treatment will include lymphodepleting chemotherapy followed by one dose of JCAR017 administered by intravenous (IV) injection.
  Arms: JCAR017 1-dose schedule
Biological: JCAR017 (lisocabtagene maraleucel) 2-dose schedule — Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JCAR017. During JCAR017 production, participants may receive low-dose chemotherapy for disease control. Upon product availability, participants will receive study treatment consisting of lymphodepleting chemotherapy followed by two IV doses of JCAR017.
  Arms: JCAR017 2-dose schedule (no longer accruing)

SUMMARY:
This open-label Phase 1 study will evaluate the safety, PK, and antitumor activity of modified T cells (JCAR017) administered to adult patients with relapsed or refractory B-cell NHL. The dose and schedule of JCAR017 will be evaluated and modified, as needed, for safety and antitumor activity. We will also determine how long the modified T cells stay in the patient's body and how well JCAR017 works in treating patients with non-Hodgkin's lymphoma whose disease has come back or has not responded to treatment.

DETAILED DESCRIPTION:
This is an open-label, multicenter Phase 1 study to determine the safety, pharmacokinetics (PK), and antitumor activity of JCAR017 in adult patients with relapsed or refractory diffuse large B cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), follicular lymphoma Grade 3B, and mantle cell lymphoma (MCL). This study will evaluate and refine the dose and schedule of JCAR017 to optimize safety and antitumor activity. A dose-confirmation group or groups will further evaluate the safety and efficacy of JCAR017 at the recommended regimen(s).

Upon successful generation of JCAR017 product, participants will receive treatment with one or more cycles of JCAR017 therapy. Each cycle will include lymphodepleting chemotherapy followed by one or two doses of JCAR017 administered by intravenous (IV) injection.

The follow-up period for each participant is approximately 24 months after the final JCAR017 infusion. Long-term follow-up for survival, toxicity, and viral vector safety will continue under a separate long-term follow-up protocol per health regulatory authority guidelines, currently up to 15 years after the last JCAR017 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Relapsed or refractory B-cell NHL, including

   1. DLBCL cohort (no longer enrolling): DLBCL, not otherwise specified (NOS; includes transformed DLBCL from indolent histology [tDLBCL]), high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (Swerdlow 2016), primary mediastinal B-cell lymphoma (PMBCL), and follicular lymphoma Grade 3B. Subjects must have been treated with an anthracycline and rituximab (or other CD20-targeted agent) and have relapsed or refractory disease after at least 2 lines of systemic therapy or after auto-HSCT.
   2. MCL cohort: MCL (diagnosis must be confirmed with cyclin D1 expression or evidence of t(11;14) by cytogenetics, fluorescent in situ hybridization [FISH], or PCR) with relapsed or refractory disease after at least 2 prior lines of systemic MCL therapy. Subjects must have been treated with an alkylating agent, Bruton's tyrosine kinase inhibitor (BTKi), and rituximab (or other CD20-targeted agent).
3. PET-positive disease by Lugano classification
4. Archived tumor biopsy tissue available from the last relapse and corresponding pathology report available or, if at least one tumor-involved site is deemed accessible at time of screening, willing to undergo pre-treatment biopsy (excisional when possible) for disease confirmation. If a subject has never had a complete response, a sample from the most recent biopsy is acceptable.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate bone marrow, renal, hepatic, pulmonary, and cardiac function
7. Adequate vascular access for leukapheresis procedure
8. Participants who have received previous CD19-targeted therapy must have CD19-positive lymphoma confirmed on a biopsy since completing the prior CD19-targeted therapy.
9. Participants must agree to use appropriate contraception.

Exclusion Criteria:

1. Active central nervous system (CNS)-only involvement by malignancy (note: participants with secondary CNS involvement are allowed on study)
2. History of other primary malignancy not in remission for at least 2 years (The following are exempt from the 2-year limit: nonmelanoma skin cancer, definitively treated stage 1 solid tumor with low risk for recurrence, curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear)
3. Treatment with alemtuzumab within 6 months of leukapheresis or fludarabine or cladribine within 3 months of leukapheresis
4. Active hepatitis B, hepatitis C, or Subjects with a history of or active human immunodeficiency virus (HIV) infectionare excluded. Subjects with active hepatitis B, or active hepatitis C are also excluded. Subjects with a negative PCR assay for viral load for hepatitis B or C are permitted. Subjects positive for hepatitis B surface antigen and/or anti-hepatitis B core antibody with negative viral load are eligible and should be considered for prophylactic antiviral therapy
5. Uncontrolled systemic fungal, bacterial, viral, or other infection
6. Presence of graft-vs-host disease (GVHD)
7. History of cardiovascular disease
8. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
9. Pregnant or nursing women
10. Use of the following:

    * Therapeutic doses of corticosteroids (defined as >20 mg/day prednisone or equivalent) within 7 days of leukapheresis or 72 hours prior to JCAR017 administration. Physiologic replacement, topical, and inhaled steroids are permitted.
    * Low dose chemotherapy (e.g., vincristine, rituximab, cyclophosphamide ≤300 mg/m2) given after leukapheresis to maintain disease control must be stopped ≥7 days prior to lymphodepleting chemotherapy.
    * Cytotoxic chemotherapeutic agents that are not considered lymphotoxic (see below) within 1 week of leukapheresis. Oral chemotherapeutic agents, including lenalidomide and ibrutinib, are allowed if at least 3 half-lives have elapsed prior to leukapheresis.
    * Lymphotoxic chemotherapeutic agents (e.g., cyclophosphamide, ifosfamide, bendamustine) within 2 weeks of leukapheresis.
    * Experimental agents within 4 weeks of leukapheresis unless no response or disease progression is documented on the experimental therapy and at least 3 half-lives have elapsed prior to leukapheresis
    * Immunosuppressive therapies within 4 weeks of leukapheresis and JCAR017 administration (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolyate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti IL6, or anti-IL6R)
    * Donor lymphocyte infusions (DLI) within 6 weeks of JCAR017 administration
    * Radiation within 6 weeks of leukapheresis. Subjects must have progressive disease in irradiated lesions or have additional non-irradiated, PET-positive lesions to be eligible. Radiation to a single lesion, if additional non-irradiated PET-positive lesions are present, is allowed up to 2 weeks prior to leukapheresis.
    * Allo-HSCT within 90 days of leukapheresis
11. Prior CAR T-cell or other genetically-modified T-cell therapy, with the exception of prior JCAR017 treatment in this protocol for subjects receiving retreatment
12. Progressive vascular tumor invasion, thrombosis, or embolism
13. Venous thrombosis or embolism not managed on a stable regimen of anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events (AEs) as assessed by CTCAE v4.03 | Up to 730 days after the final JCAR017 infusion
  Physiological parameter
Dose-limiting toxicities of JCAR017 | 28 days after first (single-dose schedule) or second (2-dose schedule) JCAR017 infusion
  Physiological parameter
Objective response rate (ORR) | 24 months
  Lugano criteria

SECONDARY OUTCOMES:
Complete response (CR) rate | 24 months
  Lugano criteria
Duration of response | 24 months
  Lugano criteria
Progression-free survival (PFS) | 24 months
  Lugano criteria
Overall survival | Up to 15 years
  Physiological parameter
Health-related quality of life | 24 months
  Questionnaire
Maximum concentration of JCAR017 (Cmax) in the peripheral blood | Up to 365 days after the final JCAR017 infusion
  qPCR
Time to maximum concentration of JCAR017 (Tmax) in the peripheral blood | Up to 365 days after the final JCAR017 infusion
  qPCR
Area-under-the-concentration-vs-time-curve (AUC) in the peripheral blood | Up to 365 days after the final JCAR017 infusion
  qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Local Institution - 0006, Birmingham, Alabama
  - Local Institution - 0007, Duarte, California
  - Local Institution - 0010, San Francisco, California
  - Local Institution - 0020, Aurora, Colorado
  - Local Institution - 0019, Atlanta, Georgia
  - Local Institution - 0003, Chicago, Illinois
  - Local Institution - 0005, Boston, Massachusetts
  - Local Institution - 0015, Boston, Massachusetts
  - Local Institution - 0008, Omaha, Nebraska
  - Local Institution - 0001, New York, New York
  - Local Institution - 0021, Charlotte, North Carolina
  - Local Institution - 0029, Pittsburgh, Pennsylvania
  - Local Institution - 0002, Houston, Texas
  - Local Institution - 0018, Seattle, Washington

REFERENCES:
- [Derived] Wang M, Siddiqi T, Gordon LI, Kamdar M, Lunning M, Hirayama AV, Abramson JS, Arnason J, Ghosh N, Mehta A, Andreadis C, Solomon SR, Kostic A, Dehner C, Espinola R, Peng L, Ogasawara K, Chattin A, Eliason L, Palomba ML. Lisocabtagene Maraleucel in Relapsed/Refractory Mantle Cell Lymphoma: Primary Analysis of the Mantle Cell Lymphoma Cohort From TRANSCEND NHL 001, a Phase I Multicenter Seamless Design Study. J Clin Oncol. 2024 Apr 1;42(10):1146-1157. doi: 10.1200/JCO.23.02214. Epub 2023 Dec 10. PMID 38072625
- [Derived] Abramson JS, Palomba ML, Gordon LI, Lunning M, Wang M, Arnason J, Purev E, Maloney DG, Andreadis C, Sehgal A, Solomon SR, Ghosh N, Dehner C, Kim Y, Ogasawara K, Kostic A, Siddiqi T. Two-year follow-up of lisocabtagene maraleucel in relapsed or refractory large B-cell lymphoma in TRANSCEND NHL 001. Blood. 2024 Feb 1;143(5):404-416. doi: 10.1182/blood.2023020854. PMID 37890149
- [Derived] Van Le H, Van Naarden Braun K, Nowakowski GS, Sermer D, Radford J, Townsend W, Ghesquieres H, Menne T, Porpaczy E, Fox CP, Schusterbauer C, Liu FF, Yue L, De Benedetti M, Hasskarl J. Use of a real-world synthetic control arm for direct comparison of lisocabtagene maraleucel and conventional therapy in relapsed/refractory large B-cell lymphoma. Leuk Lymphoma. 2023 Mar;64(3):573-585. doi: 10.1080/10428194.2022.2160200. Epub 2023 Feb 8. PMID 36755418
- [Derived] Teoh J, Brown LF. Developing lisocabtagene maraleucel chimeric antigen receptor T-cell manufacturing for improved process, product quality and consistency across CD19+ hematologic indications. Cytotherapy. 2022 Sep;24(9):962-973. doi: 10.1016/j.jcyt.2022.03.013. Epub 2022 May 21. PMID 35610089
- [Derived] Cartron G, Fox CP, Liu FF, Kostic A, Hasskarl J, Li D, Bonner A, Zhang Y, Maloney DG, Kuruvilla J. Matching-adjusted indirect treatment comparison of chimeric antigen receptor T-cell therapies for third-line or later treatment of relapsed or refractory large B-cell lymphoma: lisocabtagene maraleucel versus tisagenlecleucel. Exp Hematol Oncol. 2022 Mar 25;11(1):17. doi: 10.1186/s40164-022-00268-z. PMID 35337365
- [Derived] Ogasawara K, Lymp J, Mack T, Dell'Aringa J, Huang CP, Smith J, Peiser L, Kostic A. In Vivo Cellular Expansion of Lisocabtagene Maraleucel and Association With Efficacy and Safety in Relapsed/Refractory Large B-Cell Lymphoma. Clin Pharmacol Ther. 2022 Jul;112(1):81-89. doi: 10.1002/cpt.2561. Epub 2022 Mar 20. PMID 35156195
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Maloney DG, Kuruvilla J, Liu FF, Kostic A, Kim Y, Bonner A, Zhang Y, Fox CP, Cartron G. Matching-adjusted indirect treatment comparison of liso-cel versus axi-cel in relapsed or refractory large B cell lymphoma. J Hematol Oncol. 2021 Sep 8;14(1):140. doi: 10.1186/s13045-021-01144-9. PMID 34493319
- [Derived] Westin JR, Kersten MJ, Salles G, Abramson JS, Schuster SJ, Locke FL, Andreadis C. Efficacy and safety of CD19-directed CAR-T cell therapies in patients with relapsed/refractory aggressive B-cell lymphomas: Observations from the JULIET, ZUMA-1, and TRANSCEND trials. Am J Hematol. 2021 Oct 1;96(10):1295-1312. doi: 10.1002/ajh.26301. Epub 2021 Aug 13. PMID 34310745
- [Derived] Ogasawara K, Dodds M, Mack T, Lymp J, Dell'Aringa J, Smith J. Population Cellular Kinetics of Lisocabtagene Maraleucel, an Autologous CD19-Directed Chimeric Antigen Receptor T-Cell Product, in Patients with Relapsed/Refractory Large B-Cell Lymphoma. Clin Pharmacokinet. 2021 Dec;60(12):1621-1633. doi: 10.1007/s40262-021-01039-5. Epub 2021 Jun 14. PMID 34125421
- [Derived] Salles G, Spin P, Liu FF, Garcia J, Kim Y, Hasskarl J. Indirect Treatment Comparison of Liso-Cel vs. Salvage Chemotherapy in Diffuse Large B-Cell Lymphoma: TRANSCEND vs. SCHOLAR-1. Adv Ther. 2021 Jun;38(6):3266-3280. doi: 10.1007/s12325-021-01756-0. Epub 2021 May 10. PMID 33970454
- [Derived] Patrick DL, Powers A, Jun MP, Kim Y, Garcia J, Dehner C, Maloney DG. Effect of lisocabtagene maraleucel on HRQoL and symptom severity in relapsed/refractory large B-cell lymphoma. Blood Adv. 2021 Apr 27;5(8):2245-2255. doi: 10.1182/bloodadvances.2020003503. PMID 33904895
- [Derived] Abramson JS, Siddiqi T, Garcia J, Dehner C, Kim Y, Nguyen A, Snyder S, McGarvey N, Gitlin M, Pelletier C, Jun MP. Cytokine release syndrome and neurological event costs in lisocabtagene maraleucel-treated patients in the TRANSCEND NHL 001 trial. Blood Adv. 2021 Mar 23;5(6):1695-1705. doi: 10.1182/bloodadvances.2020003531. PMID 33720336
- [Derived] Abramson JS, Palomba ML, Gordon LI, Lunning MA, Wang M, Arnason J, Mehta A, Purev E, Maloney DG, Andreadis C, Sehgal A, Solomon SR, Ghosh N, Albertson TM, Garcia J, Kostic A, Mallaney M, Ogasawara K, Newhall K, Kim Y, Li D, Siddiqi T. Lisocabtagene maraleucel for patients with relapsed or refractory large B-cell lymphomas (TRANSCEND NHL 001): a multicentre seamless design study. Lancet. 2020 Sep 19;396(10254):839-852. doi: 10.1016/S0140-6736(20)31366-0. Epub 2020 Sep 1. PMID 32888407
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome